CLINICAL TRIAL: NCT04017065
Title: Prospective Multicenter Registry for Use of the MAXFRAME™ Multiaxial Correction System
Status: Terminated | Type: Observational
Why Stopped: Decision by the sponsor
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: MAXFRAME
Record Dates: First submitted 2019-04-17; First posted 2019-07-12 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2020-08

CONDITIONS: Limb Deformities Congenital; Limb Deformities Nos (Acquired); Deformity of Bone
Keywords: limb deformity correction; limb lengthening; MAXFRAME system
MeSH Terms: conditions — Limb Deformities, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients treated with the MAXFRAMETM system: Any patient undergoing surgical treatment (primary or revision) for deformity correction using the MAXFRAME™ system
  Interventions: Device: DePuy Synthes MAXFRAMETM system

INTERVENTIONS:
Device: DePuy Synthes MAXFRAMETM system — Patients treated with the MAXFRAMETM system will be followed up from before the surgery until the removal of the device. All treatments are based on individual clinician's judgement and the patient characteristics. The registry does not dictate any specific treatment.

SUMMARY:
The aim of this international, prospective, multicenter case series (patient registry) is to gather the first evidence on the use of the MAXFRAME™ system in normal clinical settings during deformity correction of both, the upper and lower limb, and gain information on indications, the handling of the device from the patients' and surgeons' perspective, as well as number of re-planning needed.

It is planned to prospectively follow up to 100 patients treated with the MAXFRAME™ system. Information on patients entered into the registry will be collected from before the surgery until the removal of the device.

DETAILED DESCRIPTION:
The newly developed MAXFRAME™ system from DePuy Synthes® is a multi-Axial correction system based on the hexapod configuration. The indications for the MAXFRAME™ include, but are not limited to, the treatment of open or closed fractures of long bones, pseudarthrosis, limb lengthening via epiphyseal or metaphyseal distraction, joint arthrodesis, to bridge infected fractures or non-unions, to correct bony or soft tissue deformities, and to correct of segmental defects. One of the main novelties of this system is the Perspective Frame Matching (PFM) technique. This software system uses the post-operative x-rays with the entire frame mounted to the bone to generate a 3D visualization of the frame and the exact mounting parameters as well as a representation of the deformity with regards to the position within the frame. This system generates a treatment plan according to the exact representation of the frame, and the deformity at the starting point of the correction. The risk of a frame mal-positioning is reduced, which in return is believed to reduce the risk of a false correction and hopefully leads to a more precise result. Further, this reduces the need for adaptations to the initial treatment protocol, which require repeated radiological assessment and may alienate the patient during the whole process of the deformity correction.

To the investigator's knowledge there are no published studies investigating the accuracy of this method, therefore the aim of the proposed prospective multicenter registry is to gather first evidence on the use of the MAXFRAME™ system in clinical settings and gain information on indications, handling, the number of re-planning's needed, and treatment related adverse events.

Up to 100 patients treated with the MAXFRAME™ system are planned to be included for two years enrollment period. Each patient will be followed up from before the surgery until the removal of the device.

All follow-up visits are according to standard of care. There are fixed time points (visits) during a normal deformity correction process and follow-up:

* Baseline = pre-operative assessment
* Surgery = application of the frame (defined as day 0)
* Post-OP = post-operative image assessment (for PFM planning)
* Frame removal (including conversion, if applicable)

Further, there are additional time points (visits). An additional visit is defined as every consultation during the deformity correction process, until the frame is removed, when a registry specific event of interest occurs. The events of interest for additional visits are the following:

* Re-plannings
* Re-operation / surgical interventions
* Changes to the frame
* Treatment related adverse event
* Deformity corrected

Following data points will be collected pre-, intra- and post-operatively:

Patients demographics, medical history and underlying diseases, Indication for the use of the MAXFRAMETM system, Treatment goal(s), Treatment planning, Surgical details, Changes in treatment plan, Frame removal, Radiological and calculated outcome assessment of the deformity correction and/or lengthening, Treatment-related Adverse Events, Experience with MAXFRAMETM system.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing surgical treatment (primary or revision) for deformity correction using the MAXFRAME™ system
* Informed consent obtained, i.e.:

  * Ability to understand the content of the patient information/ICF
  * Willingness and ability to participate in the clinical investigation according to the Registry Plan (RP)
  * Signed and dated IRB/EC-approved written informed consent OR
  * Written consent provided according to defined and IRB/EC approved procedures for patients who are not able to provide independent written informed consent

Exclusion Criteria:

* Participation in any other medical device or medicinal product study within the previous month that could influence the treatment observed in this registry
* Pregnancy
* Intraoperative decision to use another device than MAXFRAMETM

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patients treated with the MAXFRAMETM system for congenital or acquired deformity correction.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Baseline characteristics | baseline until the removal of the device (standard approximately 6 months)
  Demographics, medical history
Type of surgery | Day of surgery until removal of the device (standard approximately 6 months)
  primary or revision surgery
Bone lengthening measurement | baseline until the removal of the device (standard approximately 6 months)
  Bone lengthening (in mm)
Varus or valgus correction assessment | baseline until the removal of the device (standard approximately 6 months)
  Varus or valgus correction (in degrees)
Rotational correction assessment | baseline until the removal of the device (standard approximately 6 months)
  Rotational correction (in degrees)
Ante- or retro-curvature correction assessment | baseline until the removal of the device (standard approximately 6 months)
  Ante- or retro-curvature correction (in degrees)
Bone union / fusion assessment | removal of the device (standard approximately 6 months)
  Bone union / fusion (in the case of an arthrodesis)
Radiological assessments | baseline until the removal of the device (standard approximately 6 months)
  Radiological assessment according to the measured anatomical angles (degree)
Radiological assessments of deformity parameters | baseline until the removal of the device (standard approximately 6 months)
  deformity parameters depending on the level of the deformity (degree)
Reason for changes of treatment plan | baseline until the removal of the device (standard approximately 6 months)
  reason for any treatment plan changes
End of deformity correction | baseline until the removal of the device (standard approximately 6 months)
  Length gained (real (mm) according to the lengthened bone)
Assessment of the surgeon and patients experience with the MAXFRAME™ system | removal of the device (standard approximately 6 months)
  Survey with four questions to rate via numeric rating scale (0= not satisfied at all ; 10= totally satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Theodor F. Slongo, MD, Principal Investigator — University of Berne Children's Hospital Department of pediatric surgery
Locations (2):
- Penn State Hershey Bone and Joint Institute, Hershey, Pennsylvania, United States
- University of Berne Children's Hospital Department of pediatric surgery, Bern, Schweiz, Switzerland